CLINICAL TRIAL: NCT02444741
Title: Phase I/II Trial of MK-3475 and Hypofractionated Stereotactic Radiation Therapy in Patients With NSCLC
Brief Title: Pembrolizumab and Stereotactic Body Radiation Therapy or Non-Stereotactic Wide-Field Radiation Therapy in Treating Patients With Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-1020; NCI-2015-01505 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-1020 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-05-12; First posted 2015-05-14 (Estimated); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Malignant Solid Neoplasm; Metastatic Lung Non-Small Cell Carcinoma; Stage IV Lung Non-Small Cell Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated; pembrolizumab; Proton Therapy; Protons; Radiotherapy; Radiation; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Group I, Phase I (pembrolizumab + SBRT) (Experimental): Patients who exhibit a lung lesion of size and location amenable to SBRT receive pembrolizumab IV over 30 minutes on day 1. Patients also receive SBRT in 4 fractions daily on days 2-5 or either IMRT, PBRT, or 3D-CRT in 15 fractions total concurrent with pembrolizumab administration on days 1-19. Treatment repeats every 21 days for up to 16 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Radiation: Proton Beam Radiation Therapy; Radiation: Stereotactic Body Radiation Therapy
- Group I, Phase II (pembrolizumab + SBRT) (Experimental): Patients who exhibit a lung lesion with size and location amenable to SBRT receive pembrolizumab IV on day 1 and SBRT on days 44-47 or IMRT, PBT, or 3D-CRT on days 43-61. Treatment with pembrolizumab repeats every 21 days for up to 16 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Radiation: Stereotactic Body Radiation Therapy
- Group II, Phase I (pembrolizumab + IMRT, PBRT or 3D-CRT) (Experimental): Patients who exhibit a lung lesion of size or location not amenable to SBRT, but amenable to WFRT receive pembrolizumab as in Group I and either IMRT, PBRT, or 3D-CRT in 15 fractions total on days 1-19 concurrent with pembrolizumab administration.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Radiation: Proton Beam Radiation Therapy
- Group II, Phase II (pembrolizumab + XRT upon PD) (Experimental): Patients who exhibit a lung lesion with size and location amenable to SBRT receive pembrolizumab IV as in Group I without XRT. At the first planned efficacy evaluation (5 weeks), patients exhibiting PD are treated with SBRT concurrent with the remaining cycles of pembrolizumab. In the event that lesion size has progressed to the point where the attending physician no longer considers SBRT safe, then the patient will be salvaged with IMRT, PBRT, or 3D-CRT and analyzed as part of the fourth treatment group.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Radiation: Proton Beam Radiation Therapy; Radiation: Stereotactic Body Radiation Therapy
- Group III, Phase II (pembrolizumab + IMRT, PBRT, or 3D-CRT) (Experimental): Patients who exhibit a lung lesion with size and location not amenable to SBRT, but amenable to WFRT receive pembrolizumab IV as in Group I and IMRT, PBRT, or 3D-CRT on days 43-61.
  Interventions: Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Radiation: Proton Beam Radiation Therapy
- Group IV, Phase II (pembrolizumab + XRT upon PD) (Experimental): Patients who exhibit a lung lesion with size and location not amenable to SBRT, but amenable to WFRT receive pembrolizumab IV as in Group I without XRT. The decision on when to start XRT will be assessed first at week 5 (after the second dose of pembrolizumab). If a patient has PD based on irRC then XRT will be delivered after the third dose of pembrolizumab, while patients with SD or PR will not start XRT and will continue to be followed. These patients will then have follow up CT scans 5 weeks after course 3 and then approximately every 3 months for the remainder of the trial; any patient at this point with PD will then have XRT delivered with the sixth dose of pembrolizumab.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Radiation: Proton Beam Radiation Therapy
- Group V, Phase II (low dose radiation therapy) (Experimental): Patients with lesions amenable to SBRT or WFRT receive pembrolizumab IV as in Group I. Patients also receive either IMRT, PBRT, or 3D-CRT in 15 fractions to the primary lesions and low dose radiation therapy to other lesions on days 43-61 or SBRT in 4 fractions to primary lesions and low dose radiation therapy to other lesions on days 44-47.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Radiation: Proton Beam Radiation Therapy; Radiation: Radiation Therapy; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Radiation: 3-Dimensional Conformal Radiation Therapy — Undergo 3D-CRT
  Other Names: 3-dimensional radiation therapy; 3D Conformal; 3D CONFORMAL RADIATION THERAPY; 3D CRT; 3D-CRT; Conformal Therapy; Radiation Conformal Therapy; Radiation, 3D Conformal
  Arms: Group I, Phase I (pembrolizumab + SBRT); Group II, Phase I (pembrolizumab + IMRT, PBRT or 3D-CRT); Group II, Phase II (pembrolizumab + XRT upon PD); Group IV, Phase II (pembrolizumab + XRT upon PD); Group V, Phase II (low dose radiation therapy)
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
  Arms: Group I, Phase I (pembrolizumab + SBRT); Group II, Phase I (pembrolizumab + IMRT, PBRT or 3D-CRT); Group II, Phase II (pembrolizumab + XRT upon PD); Group III, Phase II (pembrolizumab + IMRT, PBRT, or 3D-CRT); Group IV, Phase II (pembrolizumab + XRT upon PD); Group V, Phase II (low dose radiation therapy)
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Radiation: Proton Beam Radiation Therapy — Undergo PBRT
  Other Names: PBRT; Proton; Proton Radiation Therapy; Radiation, Proton Beam
  Arms: Group I, Phase I (pembrolizumab + SBRT); Group II, Phase I (pembrolizumab + IMRT, PBRT or 3D-CRT); Group II, Phase II (pembrolizumab + XRT upon PD); Group III, Phase II (pembrolizumab + IMRT, PBRT, or 3D-CRT); Group IV, Phase II (pembrolizumab + XRT upon PD); Group V, Phase II (low dose radiation therapy)
Radiation: Radiation Therapy — Undergo low dose radiation therapy
  Other Names: Cancer Radiotherapy; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: Group V, Phase II (low dose radiation therapy)
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy
  Arms: Group I, Phase I (pembrolizumab + SBRT); Group I, Phase II (pembrolizumab + SBRT); Group II, Phase II (pembrolizumab + XRT upon PD); Group V, Phase II (low dose radiation therapy)

SUMMARY:
This randomized phase I/II trial studies the side effects and best dose of pembrolizumab when given together with stereotactic body radiation therapy or non-stereotactic wide-field radiation therapy (conventional radiation therapy) and to see how well they work in treating patients with non-small cell lung cancer. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Radiation therapy uses high-energy x-rays to kill tumor cells and shrink tumors. Stereotactic body radiation therapy uses special equipment to position a patient and deliver radiation to tumors with high precision. This method can kill tumor cells with fewer doses over a shorter period and cause less damage to normal tissue. Giving pembrolizumab together with radiation therapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and toxicity profile of intravenous MK-3475 (pembrolizumab) administered in combination with stereotactic body radiation therapy (SBRT) targeting 1-4 liver or thoracic lesion(s) in patients with metastatic non-small cell lung cancer (NSCLC). (Phase I) II. To evaluate the safety and toxicity profile of intravenous MK-3475 administered in combination with non-stereotactic wide-field radiation therapy (WFRT) targeting 1-4 liver or thoracic lesion(s) in patients with metastatic NSCLC. (Phase I) III. To determine the maximum tolerated dose (MTD) and dose limiting toxicities (DLTs) of MK-3475 and SBRT combination therapy. (Phase I) IV. To determine the maximum tolerated dose (MTD) and dose limiting toxicities (DLTs) of MK-3475 and WFRT combination therapy. (Phase I) V. To determine the rate of out-of-field objective responses (either complete response [CR] or partial response [PR]) of the non-irradiated disease sites. (Phase II)

SECONDARY OBJECTIVE:

I. To determine whether the addition of radiation therapy (XRT) to MK-3475 can improve the progression free survival (PFS) rate compared to MK-3475 alone. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of pembrolizumab followed by a phase II study.

PHASE I: Patients are assigned to 1 of 2 treatment groups.

GROUP I: Patients who exhibit a lung lesion of size and location amenable to SBRT receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Patients also receive SBRT in 4 fractions daily on days 2-5 or either intensity modulated radiation therapy (IMRT), proton beam radiation therapy (PBRT), or 3 dimensional conformation radiation therapy (3D-CRT) in 15 fractions total concurrent with pembrolizumab administration on days 1-19. Treatment repeats every 21 days for up to 16 courses in the absence of disease progression or unacceptable toxicity.

GROUP II: Patients who exhibit a lung lesion of size or location not amenable to SBRT, but amenable to WFRT receive pembrolizumab as in Group I and either IMRT, PBRT, or 3D-CRT in 15 fractions total concurrent with pembrolizumab administration.

PHASE II: Patients for whom SBRT is recommended are randomized to Group 1 or 2, patients for whom conventional radiation therapy is recommended are randomized to Group 3 or 4, and patients with lesions amenable to SBRT or WFRT are assigned to Group 5.

GROUP I: Patients who exhibit a lung lesion with size and location amenable to SBRT receive pembrolizumab IV on day 1 and SBRT on days 44-47 or IMRT, PBT, or 3D-CRT on days 43-61. Treatment with pembrolizumab repeats every 21 days for up to 16 courses in the absence of disease progression or unacceptable toxicity.

GROUP II: Patients who exhibit a lung lesion with size and location amenable to SBRT receive pembrolizumab IV as in Group I without XRT. At the first planned efficacy evaluation (5 weeks), patients exhibiting progressive disease (PD) are treated with SBRT concurrent with the remaining cycles of pembrolizumab. In the event that lesion size has progressed to the point where the attending physician no longer considers SBRT safe, then the patient will be salvaged with IMRT, PBRT, or 3D-CRT and analyzed as part of the fourth treatment group.

GROUP III: Patients who exhibit a lung lesion with size and location not amenable to SBRT, but amenable to WFRT receive pembrolizumab IV as in Group I and IMRT, PBRT, or 3D-CRT on days 43-61.

GROUP IV: Patients who exhibit a lung lesion with size and location not amenable to SBRT, but amenable to WFRT receive pembrolizumab IV as in Group I without XRT. The decision on when to start XRT will be assessed first at week 5 (after the second dose of pembrolizumab). If a patient has PD based on immune response related criteria (irRC) then XRT will be delivered after the third dose of pembrolizumab, while patients with stable disease (SD) or PR will not start XRT and will continue to be followed. These patients will then have follow up computed tomography (CT) scans 5 weeks after course 3 three and then approximately every 3 months for the remainder of the trial; any patient at this point with PD will then have XRT delivered with the sixth dose of pembrolizumab.

GROUP V: Patients with lesions amenable to SBRT or WFRT receive pembrolizumab IV as in Group I. Patients also receive either IMRT, PBRT, or 3D-CRT in 15 fractions to the primary lesions and low dose radiation therapy to other lesions on days 43-61 or SBRT in 4 fractions to primary lesions and low dose radiation therapy to other lesions on days 44-47.

After completion of study treatment, patients are followed up at 30 days and then every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed non-small lung cancer; for patients in group 5, any solid tumor histology to be included
* Stage IV metastatic disease (only during the phase II)
* At least one thoracic or liver lesion amenable to radiation, for group 5 we need one area that can safely receive SBRT or WFRT, not restricted to lung or liver sites
* At least one additional non-contiguous lesion to the irradiated lesion amenable to radiographic evaluation
* Be willing and able to provide written informed consent/assent for the trial
* Have measurable disease based on immune related response criteria (irRC) criteria
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Absolute neutrophil count (ANC) >= 1,500 /mcL (performed within 28 days prior to study registration up to the first dose of study drug)
* Platelets >= 100,000 /mcL (performed within 28 days prior to study registration up to the first dose of study drug)
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L (performed within 28 days prior to study registration up to the first dose of study drug)
* Serum creatinine =< 1.5 X upper limit of normal (ULN) or measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or calculated creatinine clearance [CrCl]) or >= 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN (creatinine clearance should be calculated per institutional standard) (performed within 28 days prior to study registration up to the first dose of study drug)
* Serum total bilirubin =< 1.5 X ULN or direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN (performed within 28 days prior to study registration up to the first dose of study drug)
* Aspartate aminotransferase (AST) serum glutamic-oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT) serum glutamic-pyruvic transaminase (SGPT) =< 2.5 X ULN or =< 5 X ULN for subjects with liver metastases (performed within 28 days prior to study registration up to the first dose of study drug)
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or partial prothrombin time (PTT) is within therapeutic range of intended use of anticoagulants (performed within 28 days prior to study registration up to the first dose of study drug)
* Activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants (performed within 28 days prior to study registration up to the first dose of study drug)
* Patients with brain metastasis will be included as long as they are free of neurologic symptoms related to metastatic brain lesions and who do not require or receive systemic corticosteroid therapy in the 14 days prior to beginning MK-3475 therapy
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication; subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy
* We will allow XRT prior to study entry to other sites, with no washout period, allowed prior to study entry as long as at least one measurable sites of disease is kept unirradiated

Exclusion Criteria:

* Is currently participating in or has participated in a study of an investigational agent (except glutamine) or using an investigational device within 4 weeks of the first dose of treatment or 5 half lives, whichever is shorter
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment; unless the steroid therapy is for physiological replacement
* Has a diagnosis of active scleroderma, lupus, or other autoimmune disease which by the opinion of the treating radiation oncologist precludes safe radiation therapy
* Has had prior radiation therapy to all available thoracic and liver lesions such that additional radiation therapy is unsafe by the opinion of the treating radiation oncologist
* Has had a prior monoclonal antibody within 4 weeks or 5 half-lives, which ever is shorter, prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Has had prior chemotherapy or targeted small molecule therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent

  * Note: Subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study
  * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis; subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment
* Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents; subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule; subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study; subjects with hypothyroidism stable on hormone replacement or Sjogren's syndrome will not be excluded from the study
* Has evidence of interstitial lung disease or active, non-infectious pneumonitis
* Has an active infection requiring systemic therapy or hospital admission
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B virus HBsAg surface protein antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has received a live vaccine within 30 days prior to the first dose of trial treatment
* Symptomatic brain metastasis
* Has experienced a dose limiting toxicity on treatment with either prior radiation or anti programmed cell death 1 (PD-1) or programmed cell death 1 ligand 1 (PD-L1) inhibitor therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2015-09-17 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Disease response, according to immune related response criteria (Phase I/II) | Beginning 3 months after initiation of treatment
  Treatment success will be defined as radiographic complete response or partial response measured using Pearson chi-squared or Fisher exact tests.
Incidence of toxicity (Phase I/II) | Up to 90 days after completion of treatment
  Graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0.
Maximum tolerated dose of pembrolizumab and stereotactic body radiation therapy (Phase I) | 22 days
  Graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0.
Maximum tolerated dose of pembrolizumab and non-stereotactic wide-field radiation therapy (Phase I) | 22 days
  Graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0.
Objective response (complete response + partial response) of the non-irradiated disease sites, according to Out-Field immune related response criteria (Phase II) | Up to 5 years
  Assesed according to Out-Field immune related response criteria. Treatment success will be defined as radiographic complete response or partial response measured using Pearson chi-squared or Fisher exact tests.

SECONDARY OUTCOMES:
Progression-free survival (Phase II) | From the time of enrollment to first evidence of progressive disease, assessed at 3 months after treatment initiation
  Analysis conducted using Kaplan-Meier method. At the discretion of the investigators, multivariate Cox regression will be done to adjust for (among other factors): number of metastatic disease sites, number of prior treatments, primary cancer histology, age, pre-treatment Karnofsky performance scale, and Royal Marsden score.
Overall survival | Receipt of the first pembrolizumab dose to death, assessed up to 5 years
  Analysis conducted using Kaplan-Meier method, with comparisons regarding overall survival made via the log-rank test. At the discretion of the investigators, multivariate Cox regression will be done to adjust for (among other factors): number of metastatic disease sites, number of prior treatments, primary cancer histology, age, pre-treatment Karnofsky performance scale, and Royal Marsden score.

CONTACTS AND LOCATIONS:
Overall Officials: James Welsh, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Butner JD, Martin GV, Wang Z, Corradetti B, Ferrari M, Esnaola N, Chung C, Hong DS, Welsh JW, Hasegawa N, Mittendorf EA, Curley SA, Chen SH, Pan PY, Libutti SK, Ganesan S, Sidman RL, Pasqualini R, Arap W, Koay EJ, Cristini V. Early prediction of clinical response to checkpoint inhibitor therapy in human solid tumors through mathematical modeling. Elife. 2021 Nov 9;10:e70130. doi: 10.7554/eLife.70130. PMID 34749885
- [Derived] Theelen WSME, Chen D, Verma V, Hobbs BP, Peulen HMU, Aerts JGJV, Bahce I, Niemeijer ALN, Chang JY, de Groot PM, Nguyen QN, Comeaux NI, Simon GR, Skoulidis F, Lin SH, He K, Patel R, Heymach J, Baas P, Welsh JW. Pembrolizumab with or without radiotherapy for metastatic non-small-cell lung cancer: a pooled analysis of two randomised trials. Lancet Respir Med. 2021 May;9(5):467-475. doi: 10.1016/S2213-2600(20)30391-X. Epub 2020 Oct 20. PMID 33096027
- [Derived] Welsh J, Menon H, Chen D, Verma V, Tang C, Altan M, Hess K, de Groot P, Nguyen QN, Varghese R, Comeaux NI, Simon G, Skoulidis F, Chang JY, Papdimitrakopoulou V, Lin SH, Heymach JV. Pembrolizumab with or without radiation therapy for metastatic non-small cell lung cancer: a randomized phase I/II trial. J Immunother Cancer. 2020 Oct;8(2):e001001. doi: 10.1136/jitc-2020-001001. PMID 33051340
- [Derived] Chen D, Menon H, Verma V, Guo C, Ramapriyan R, Barsoumian H, Younes A, Hu Y, Wasley M, Cortez MA, Welsh J. Response and outcomes after anti-CTLA4 versus anti-PD1 combined with stereotactic body radiation therapy for metastatic non-small cell lung cancer: retrospective analysis of two single-institution prospective trials. J Immunother Cancer. 2020 Jan;8(1):e000492. doi: 10.1136/jitc-2019-000492. PMID 31996395
- See also: MD Anderson Cancer Center — http://www.mdanderson.org